CLINICAL TRIAL: NCT05316142
Title: Evaluation of the Effect of Subconjunctival 5-fluorouracil on the Outcome of Ahmed Valve in Neovascular Glaucoma: Randomized Clinical Trial
Brief Title: Effect of Subconjunctival 5-fluorouracil on the Outcome of Ahmed Valve in Neovascular Glaucoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1400-2-86-21845
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-09

CONDITIONS: Neovascular Glaucoma
Keywords: Neovascular Glaucoma (NVG); Ahmed Glaucoma Valve (AGV); 5FU; MMC
MeSH Terms: conditions — Glaucoma, Neovascular

STUDY DESIGN:
Intervention Model Description: Clinical trial study with two parallel groups, randomized using computer permuted block randomization, 35 patients in each group are included and followed up for at least 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AGV with intraoperation MMC and postoperative BSS (Active Comparator): Patients with neovascular glaucoma undergoing shunt implant surgery with MMC during surgery. This method will use Ahmad FP7 model valved shunt (New World Medical, LA), which is one of the most commonly used shunts in the world. First, MMC at a dose of 0.04% is placed in the shunt plate for two minutes and then rinsed. The shunt is fixed and then the shunt tube is inserted into the eye and fixed with nylon 10.0 thread. The conjunctiva is also swabbed with 8.0 vicryl sutures. After the operation, patients undergo regular examinations according to a specific protocol to evaluate the effectiveness as well as possible complications.
  Also in the first, third and fifth weeks, BSS injections are given as a subconjugate with a volume of 0.1 ml.
  Interventions: Procedure: AGV with intraoperation MMC and postoperative BSS
- AGV with intraoperation MMC and postoperation 5FU (Active Comparator): Patients with neovascular glaucoma undergoing shunt implant surgery with MMC during and 5FU after surgery .This method will use Ahmad FP7 model valved shunt (New World Medical, LA), which is one of the most commonly used shunts in the world. First, 5FU at a dose of 0.04% is placed in the shunt plate for two minutes and then rinsed. The shunt is fixed and then the shunt tube is inserted into the eye and fixed with nylon 10.0 thread. The conjunctiva is also swabbed with 8.0 vicryl sutures. After the operation, patients undergo regular examinations according to a specific protocol to evaluate the effectiveness as well as possible complications. Also in the first, third and fifth weeks, 5FU injections are given as a subconjugate with a volume of 0.1 ml containing 5 mg of the drug.
  Interventions: Procedure: AGV with intraoperation MMC and post operation 5FU

INTERVENTIONS:
Procedure: AGV with intraoperation MMC and postoperative BSS — This method will use Ahmad FP7 model valved shunt (New World Medical, LA), which is one of the most commonly used shunts in the world
  Arms: AGV with intraoperation MMC and postoperative BSS
Procedure: AGV with intraoperation MMC and post operation 5FU — This method will use Ahmad FP7 model valve shunt (New World Medical, LA). First, 5FU at a dose of 0.04% is placed in the shunt plate for two minutes and then rinsed.
  Arms: AGV with intraoperation MMC and postoperation 5FU

SUMMARY:
Neovascular glaucoma is a common and severe type of secondary closed-angle glaucoma. Topical treatments have variable effects and unfortunately often require surgery to control IOP. Although Glaucoma Drainage Device (GDD) such as Ahmed Glaucoma Valve (AGV) are a surgical choice in these patients, their effectiveness decreases over time.

One of the main causes of failure in AGV surgery is the formation of scar tissue and fibrosis around the shunt plate.

So, the aim of this study was to evaluate the effect of using MMC Intraoperative and 5FU Postoperative with AGV surgery in neovascular glaucoma patients according to a specific protocol, on the incidence of Hypertensive Phase (HP) and surgical success rate.

DETAILED DESCRIPTION:
All patients with neovascular glaucoma who need surgery for the first time are included in the study. Inclusion criteria include patients over 18 years of age with neovascular glaucoma whose IOP is not controlled by medical treatment. Exclusion criteria Study includes: No Light Perception patients, age less than 18 years, history of any type of eye surgery including previous glaucoma and retinal surgeries (except uncomplicated cataract surgery), history of cyclodestructive procedures, pregnant patients.

Patients after obtaining a history, especially of drugs and underlying diseases, under complete ophthalmic examination including: visual acuity (VA) and BCVA with Snelln chart, examination with slit lamp and performing dynamic gonioscopy using, IOP measurement with Goldmann Applanation Tonometer and corneal thickness measurement (CCT). . Patients are then randomized using permuted block design computer and placed in two groups of AGV surgery with anti-fibrotic treatment and AGV surgery alone.

In AGV surgery, the conjunctiva of the superotemporal area is first dissected. The plate shunt is then threaded 10 mm from the limbus to the sclera with non-absorbable proline thread. The tube insertion is then performed using a 23g needle, and after fixing the scleral patch, the conjugate is threaded with 8.0 vicryl thread and the shunt surgery is completed.

In all patients during surgery and before fixing the shunt plate, MMC is used with a sponge at a dose of 0.2 mg / ml for 2 minutes and then washed with a large amount of BSS. All patients receive intraviteral bevacizumab at the end of the operation. In the postoperative anti-fibrotic group during F/U in the first, third and fifth weeks, 5FU subconjunctival injection is performed after local anesthesia with tetracaine behind the slit lamp for all patients with a pressure above 6 mm Hg. 5FU with a volume of 0.1 ml containing 5 mg of drug is injected in the area of the tendon adjacent to the shunt plate.

After surgery, patients undergo regular examinations. Patients at least on the first day, first week, third week, fifth week, third month, sixth month, twelfth month in terms of visual acuity, refraction, IOP, various surgical complications, the number of drugs used to control IOP are evaluated.

ELIGIBILITY:
Inclusion Criteria:

• Patients with diagnosis of neovascular glaucoma

Exclusion Criteria:

* Patients with no light perception
* Patients aged less than 18 years old
* History of previous GDD implantation
* History of cyclodestructive procedures
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate (SR) | Sixth month
  1. Reduction of at least 20% IOP after surgery 2. 21> IOP> 6 with or without medication
Hypertensive Phase (HP) | Third month
  IOP>21 after surgery

SECONDARY OUTCOMES:
Number of mediaction | Sixth month
  Number of antiglauocoma medication after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Iran University of Medical Sciences, Tehran, Iran